CLINICAL TRIAL: NCT06281366
Title: Diamine Oxidase and Adverse Pregnancy Outcomes
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: DR Healthcare (Unknown)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)470-2023
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Complications
Keywords: Preeclampsia; PPROM; preterm birth; Fetal death; Low birthweight
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia; Preterm Premature Rupture of the Membranes; Premature Birth; Fetal Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Pregnant women with a positive first-trimester screening for preeclampsia (high risk) and no pregnancy complications (preeclampsia, fetal death, preterm birth, PPROM, low birthweight).
- Cases: Pregnant women with a positive first-trimester screening for preeclampsia (high risk) and any of the following pregnancy complications: preeclampsia, fetal death, preterm birth, PPROM, low birthweight.

SUMMARY:
In normal pregnancies, blood histamine concentration remains within normal values; however, the serum histaminolytic activity is increased. Histamine is mainly produced by mast cells, platelets, basophils, neurons and enterochromatin cells, where it is stored and released when required. Reduced DAO activities have been found in high-risk pregnancies. Lower DAO activity has been associated to miscarriage, fetal demise, preeclampsia, low birthweight and preterm birth. The placenta is very rich in DAO activity and is the principal source of increased histaminolytic activity in normal pregnancies.

First-trimester screening for preeclampsia (PE) is a routine screening which is performed in the first trimester. Women with a positive result are at a greater risk of PE but also other pregnancy complications such as stillbirth, preterm birth and low birthweight. These cases are prescribed aspirin until term. This intervention has demonstrated to significantly reduce the risk of PE and other complications. Unfortunately, aspirin does not avoid all cases with adverse outcomes, indicating that additional mechanisms may be involved in the development of such pregnancy complications, such as DAO decreased activity.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Maternal age ≥18
* High risk (≥1/50) in the first-trimester screening for preeclampsia
* Gestational age between 11+0 and 16+6 weeks of gestation

Exclusion Criteria:

* Fetal malformation
* Fetal death
* Maternal digestive inflammatory disease or intolerance
* Refusal to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single pregnancies between 11+0 and 16+6 weeks of gestation and high risk for preeclampsia in the first trimester screening (risk ≥1/50)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diamine oxidase activity first trimester | 11-16+6 weeks of gestation
  diamine oxidase enzime activity in maternal blood
Diamine oxidase gene polymorphisms | 11-16+6 weeks of gestation
  variants of the AOC1 gene: rs10156191, rs1049742, rs1049793 and rs2052129

SECONDARY OUTCOMES:
Blood Diamine oxidase activity at delivery | At the time of delivery
  diamine oxidase enzime activity in maternal blood
Placental Diamine oxidase activity at delivery | At the time of delivery
  diamine oxidase enzime activity in placenta
Blood histamine levels at delivery | At the time of delivery
  histamine levels in maternal blood
Placental histamine levels at delivery | At the time of delivery
  histamine levels in placenta
Urine histamine levels at delivery | At the time of delivery
  histamine levels in 24-hour maternal urine

CONTACTS AND LOCATIONS:
Locations (1):
- Manel Mendoza, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided